CLINICAL TRIAL: NCT07369206
Title: Association of Admission Syndromic Diagnoses With ICU Mortality in a Mixed Adult Intensive Care Unit: Retrospective Cohort
Brief Title: ICU Admission Diagnoses and ICU Mortality
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet Akif Yilmaz, Principal Investigator, Ataturk University
Other Study IDs: ICU-RETRO-2025; 2026/1 (Other: Atatürk University Clinical Research Ethics Committee)
Record Dates: First submitted 2026-01-08; First posted 2026-01-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Critical Illness; Sepsis; Septic Shock; Acute Respiratory Distress Syndrome (ARDS); Acute Respiratory Failure; Multiple Organ Dysfunction Syndrome
Keywords: Intensive Care Unit; ICU Mortality; Admission Diagnosis; Retrospective Cohort; Severity Score; APACHE II; SAPS; SOFA; Length of Stay
MeSH Terms: conditions — Critical Illness; Sepsis; Shock, Septic; Respiratory Distress Syndrome; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult ICU admissions (2025): Adult patients (≥18 years) admitted to a tertiary mixed intensive care unit between January 1, 2025 and December 31, 2025. For patients with multiple ICU admissions, only the first ICU admission will be included. Data will be abstracted retrospectively from electronic medical records and ICU charts; variables will be recorded based on the first 24 hours after ICU admission.

SUMMARY:
This retrospective cohort study will evaluate whether syndromic clinical diagnoses present at ICU admission are associated with ICU mortality, independent of physiologic severity scores. Adult patients admitted to a tertiary mixed ICU during 2025 will be assessed.

DETAILED DESCRIPTION:
Data will be obtained retrospectively from the hospital information system and ICU clinical records. Variables will be recorded based on the first 24 hours after ICU admission. Demographics, admission characteristics, comorbidities, severity scores (APACHE II, SAPS, SOFA), and admission syndromic diagnoses (e.g., sepsis/septic shock, acute respiratory failure, ARDS, MODS) will be collected. The primary outcome is ICU mortality; secondary outcomes include ICU length of stay and ICU discharge disposition.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) admitted to the ICU between January 1, 2025 and December 31, 2025.
* If a patient has more than one ICU admission during the study period, only the first ICU admission will be included.

Exclusion Criteria:

* ICU stay <24 hours.
* Missing essential data preventing assessment of the primary outcome (ICU mortality) and/or calculation of severity scores (APACHE II, SAPS, SOFA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the tertiary mixed ICU of Atatürk University Faculty of Medicine (Department of Anesthesiology and Reanimation) between January 1 2024 and December 31 2025. Data will be collected retrospectively from hospital information systems and ICU records, based on the first 24 hours after ICU admission.
Sampling Method: Non-Probability Sample
Enrollment: 1248 (Actual)
Dates: Start 2026-01-30 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
ICU mortality | From ICU admission until ICU discharge (end of index ICU stay), assessed up to 90 days
  Death occurring during the index ICU stay (ICU mortality), abstracted from electronic medical records.

SECONDARY OUTCOMES:
ICU length of stay (LOS) | From ICU admission to ICU discharge (index ICU stay), assessed at ICU discharge (up to 90 days)
  ICU length of stay (days) during the index ICU admission, calculated as the difference between ICU admission and ICU discharge timestamps in the electronic medical record.
ICU discharge disposition | At ICU discharge (index ICU stay; assessed at the time of ICU discharge in the medical record, up to 90 days)
  Disposition at ICU discharge categorized as: death in ICU, transfer to hospital ward, or transfer to another facility; determined from the ICU discharge documentation in the electronic medical record.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset is derived from retrospective hospital records and contains potentially identifiable information.

REFERENCES:
- [Background] Le Gall JR, Lemeshow S, Saulnier F. A new Simplified Acute Physiology Score (SAPS II) based on a European/North American multicenter study. JAMA. 1993 Dec 22-29;270(24):2957-63. doi: 10.1001/jama.270.24.2957. Erratum in: JAMA 1994 May 4;271(17):1321. PMID: 8254858.
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID: 3928249.
- [Background] Angus DC, van der Poll T. Severe sepsis and septic shock. N Engl J Med. 2013 Nov 21;369(21):2063. doi: 10.1056/NEJMc1312359. PMID: 24256390
- [Background] Vincent JL, Marshall JC, Namendys-Silva SA, François B, Martin-Loeches I, Lipman J, Reinhart K, Antonelli M, Pickkers P, Njimi H, Jimenez E, Sakr Y; ICON investigators. Assessment of the worldwide burden of critical illness: the intensive care over nations (ICON) audit. Lancet Respir Med. 2014 May;2(5):380-6. doi: 10.1016/S2213-2600(14)70061-X. Epub 2014 Apr 14. PMID: 24740011